CLINICAL TRIAL: NCT07164495
Title: Investigation of the Risk Factors and Establishing a Prediction Model for Developing Peak Foot Pressure During Walking in the Diabetic Patients
Brief Title: Risk Factors for Developing Peak Plantar Pressure During Walking in the Diabetic Patients
Status: Recruiting | Type: Observational
Sponsor: China Medical University Hospital (Other)
Collaborators: China Medical University, Taiwan (Other)
Responsible Party: Principal Investigator, Hsiu-Chen Lin, Professor, China Medical University, Taiwan
Other Study IDs: CMUH113-REC1-169
Record Dates: First submitted 2025-08-29; First posted 2025-09-10 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Diabete Type 2
Keywords: Diabetes; Gait; Plantar Pressure
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- type 2 diabetes: 1. Diagnosed with type 2 diabetes;
  2. Able to walk at least 10 meters independently without any assistive device;
  3. Age > 18 years.
  4. No acute foot ulcers, any lower limb deformity or surgery, neurological disease that may affect walking function.
  5. No Cognitive impairment and inability to follow instructions.

SUMMARY:
The goal of this observational study is to investigate the clinically convenient dynamic and static measurement parameters to identify related risk factors of developing high peak plantar pressure during walking in the type-2 diabetic patients, and then establish a predictive model to estimate the likelihood of excessive plantar pressure.

The main question it aims to answer is:

Which clinical measurements may be used as the predictors that increased peak plantar pressure in the type-2 diabetic patients? Participants taking the examinations will understand their own clinally meaningful measurements related to their plantar pressure during walking. Further thorough analysis will be employed to develop a predictive model, aiming to provide potential improvement strategies for preventing diabetic foot ulcers in the future.

DETAILED DESCRIPTION:
Diabetes is one of the top three chronic diseases among the population, with type 2 diabetes accounting for 90% of all cases. Due to decreased insulin sensitivity, the body cannot effectively store glucose in muscle, fat, and liver cells, leading to elevated blood sugar levels. This condition often results in various comorbidities and complications, with diabetic peripheral neuropathy (DPN) being the most prominent. DPN symptoms include loss of sensation to pain, pressure, vibration, proprioception, and temperature changes, which can lead to foot ulcers and altered gait in patients. The primary risk factor for diabetic foot ulcers is excessive or concentrated plantar pressure. Currently, the main preventive measure for diabetic foot ulcers is the use of insoles or footwear to reduce foot pressure. However, the difficulty in obtaining plantar pressure monitoring equipment limits its widespread clinical use. In contrast, assessments of foot morphology and range of motion (ROM), as well as the application of new sensors for gait kinematic measurement, are relatively convenient for clinical use. Therefore, this study aims to establish the relationship between peak plantar pressure during walking in diabetic patients and clinically convenient dynamic and static measurement parameters, identify related risk factors, and develop a predictive model to estimate the likelihood of excessive plantar pressure.

The study plans to recruit 120 diabetic patients, using the NDS scale to measure participants' neuropathy disability levels, Von Frey monofilaments to assess plantar sensation, goniometers to record joint angles of the first metatarsophalangeal joint, ankle, and knee, graph paper to record foot shape, RehaGait(R) gait analysis system to record walking kinematics, and Noraxon(R) Ultium Insole to record plantar pressure values. Subsequently, correlation analysis will be used to identify the relationship between joint angles, foot shape, walking kinematics, and peak plantar pressure values, while chi-square tests will identify significant risk factors. Finally, multiple regression analysis will be employed to develop a predictive model, aiming to provide potential improvement strategies for preventing diabetic foot ulcers in the future.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with type 2 diabetes, at least for five years
* aged older than 18 years
* walk independently for at least 10 meter without any assistive device

Exclusion Criteria:

* severe deformity in the foot or lower extremity
* significant neuropathic or surgical diseases that affect normal walking function
* cognitive dysfunction
* active foot ulcer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: those diagnosed with type 2 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
plantar pressure | Day 1: a single time point
  Pressure insole will be inserted into the standard shoes to record plantar pressure values during level walking

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University, Department of Physical Therapy, Taichung, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No